CLINICAL TRIAL: NCT01285206
Title: A Study To Determine Whether Carbon Polymer Blankets Can Reduce The During And After Short, Day Operations
Brief Title: Carbon Polymer Blankets to Prevent Incidence Of Peri-Operative Hypothermia (IPH) in the DSU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brighton and Sussex University Hospitals NHS Trust (Other)
Responsible Party: Dr M Sharma, Brighton and Sussex University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10/H1107/5
Record Dates: First submitted 2011-01-25; First posted 2011-01-27 (Estimated); Last update posted 2011-01-27 (Estimated); Status verified 2010-09

CONDITIONS: Hypothermia
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Routine practice (Experimental)
  Interventions: Device: Carbon polymer warming blanket

INTERVENTIONS:
Device: Carbon polymer warming blanket — Routine practice ( + no carbon polymer blanket) versus use of HotDog carbon polymer warming blanket throughout day surgery procedure
  Other Names: HotDog warming blanket

SUMMARY:
Patients whose temperature drops below 36.0 degrees Centigrade during or after surgery suffer more complications, such as wound infections and increased blood loss, resulting in more blood transfusions and longer hospital stays than those who don't.

There is evidence that even a drop below 36.5 degrees Centigrade is sufficient to cause significant adverse effects. Although there is much evidence regarding the effectiveness of warming for long operations, there is nothing looking at short procedures such as those undertaken in the daysurgery setting.

A new carbon polymer blanket (HotDog Augustine Biomedical and Design) has been shown, in volunteer studies, to be as effective as forced air warming blankets (which are used for long operations) in preventing hypothermia. In contrast to forced air, the carbon polymer is reusable and has lower running-costs so is likely to be cheaper in the long term. This is particularly relevant in the day surgery setting where high numbers of patients are operated on. Additionally, and unlike the forced air warmers, the blanket can run on a battery so it can be applied from the moment the patient goes to sleep to the moment they wake up so it could actually prove more effective at preventing hypothermia in the clinical setting. This study aims to determine whether the carbon polymer blankets can reduce the incidence of hypothermia in the day surgery (ie. short operating time) setting.

DETAILED DESCRIPTION:
Recently published NICE guidelines recommend using fluid warmers for all infusions of 500mls or more and forced-air warming blankets for all main theatre operations. These guidelines have been extrapolated from work done on longer operations.

Patients whose temperature drops below 36 degrees Centigrade during or after surgery suffer more complications and blood loss than those whose temperature remains above 36 degrees Centigrade. They also often require more blood transfusions and stay in hospital for longer. Some of these complications are more common even when the temperature drops below 36.5.

Disposable forced-air warming blankets prevent hypothermia, but cannot be re-used and therefore incur a significant expense in terms of consumables.

Re-usable carbon polymer blankets, such as the HotDog, have been shown to not only be effective in preventing hypothermia, but have also been shown to maintain core temperature as effectively as forced air blankets.

Carbon polymer blankets are re-usable, with the added associated benefit of lower running costs. Therefore, in the face of limited NHS resources a reusable money saving alternative, such as the carbon polymer HotDog, would be a preferred option to the disposable forced air blanket.

The current data on the effectiveness of the carbon polymer blanket is from volunteers. This study is actually powered to show a reduction in the number of patients who get cold in a clinical setting.

References:

NICE. Perioperative hypothermia (inadvertent): the management of inadvertent peri-operative hypothermia in adults.NICE Clinical Guideline 29. London: National Institute for Health and Clinical Excellence, 2008. http://www.nice.org.uk/GC065.

Schmeid H, Kurz A, Sessler DI, Kozek S, Reiter A. Mild hypothermia increases blood loss and transfusion requirements during total hip arthroplasty. The Lancet 1996; 347:289-92.

Rajagopalan S, Mascha E, Na J, Sessler DI: The Effects of Mild Perioperative Hypothermia on Blood Loss and Transfusion Requirement. Anesthesiology 2008;108:717.

ELIGIBILITY:
Inclusion Criteria:

* All patients, who are scheduled for non-emergency daycase surgery which will take place with them in the supine position

Exclusion Criteria:

* Those patients who refuse
* Who are unable to fully understand the trial and give valid
* Informed consent; OR
* Who will not be positioned supine on the operating table

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Core temperature | Every 15 minutes
  Temperatures will be taken:
  Preoperatively on the day case unit ward, At the beginning of the operation Every 15 minutes thereafter intraoperatively. At the end of the operation in recovery Every 30 minutes until discharged home.

SECONDARY OUTCOMES:
Total blood loss | At the end of the operative procedure
  Total blood loss will be recorded by surgical team. Blood collected in suction cannister and estimated blood loss from surgical swab wet vs. dry weight
Blood transfusion | From the start of the operation until discharge. If patient is re-admitted within 24 hours requiring blood transfusion - also be counted
  Whether a blood transfusion has taken place as a direct consequence of the operation will be recorded in the patients notes. The type and amount of blood products given will also be recorded in the patients notes and by the hospital blood bank services
Wound infection | Upon patient discharge/ At GP follow-up at one month
  The development of a wound infection will either be recorded in the patient's notes if associated with the patient's hospital stay, or the information will be obtained from the GP follow-up phone-call.
Shivering (need for treatment or not) | Recorded during recovery stay
  The occurrence of shivering (andneed for treatment or not) will be recorded by the recovery staff on the questionnaire sheets
Time in recovery | Recorded during recovery stay
  This will recorded by the recovery staff as entry time and discharge time from recovery.
Time taken for patient to be considered fit for discharge i.e. length of hospital stay. | Upon discharge from hospital
  This data will be taken from the patient's notes: operation date until date of (fit for) discharge from hospital

CONTACTS AND LOCATIONS:
Overall Officials: C. Mark Harper, MBBS, Study Director — Brighton and Sussex University Hospitals NHS Trust
Locations (1):
- Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex, United Kingdom

REFERENCES:
- See also: HotDog Warming Blanket webpage link — http://www.hotdogwarming.com/